CLINICAL TRIAL: NCT05445934
Title: A Phase II/III, Double-Blind, Randomized, Placebo-controlled, Multicenter Study to Evaluate the Efficacy and Safety of FB2001 in Hospitalized Patients With Moderate to Severe COVID-19
Brief Title: Evaluate the Efficacy and Safety of FB2001 in Hospitalized Patients With Moderate to Severe COVID-19 (BRIGHT Study)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Frontier Biotechnologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FB2001-301
Record Dates: First submitted 2022-06-27; First posted 2022-07-06 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: COVID-19
Keywords: severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2)
MeSH Terms: conditions — COVID-19 | interventions — FB2001

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FB2001 group (Experimental): FB2001 will be administered by IV infusion twice daily (BID) for up to 5 days, plus SOC.
  Interventions: Drug: FB2001
- Placebo group (Placebo Comparator): Placebo will be administered by IV infusion twice daily (BID) for up to 5 days, plus SOC.
  Interventions: Drug: FB2001 placebo

INTERVENTIONS:
Drug: FB2001 — FB2001 for injection will be reconstituted with 100 mL of normal saline prior to intravenous infusion. FB2001 will be administered by IV infusion over approximately 60 minutes.
  Other Names: DC402234
  Arms: FB2001 group
Drug: FB2001 placebo — Placebo will be reconstituted with 100 mL of normal saline prior to intravenous infusion. Placebo will be administered by IV infusion over approximately 60 minutes.
  Arms: Placebo group

SUMMARY:
This study is a double-blind, randomized, placebo-controlled study to evaluate the efficacy and safety of FB2001 in hospitalized patients with moderate to severe Coronavirus Disease 2019 (COVID-19). A total of about 1188 subjects are planned to be enrolled. The subjects will be randomized in a 1:1 ratio to FB2001 group or placebo group while both receiving standard of care treatment.

DETAILED DESCRIPTION:
Coronavirus Disease 2019 (COVID-19) is a respiratory illness that can spread from person to person. The infectious agent that causes COVID 19 is a novel coronavirus, named severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), was first identified during a recent outbreak in December 2019. Patients with COVID-19 have symptoms of fever, cough, and shortness of breath along with non-specific symptoms including myalgia and fatigue.

FB2001 is a small-molecule inhibitor of coronavirus 3CL protease (3CLpro). In two phase I clinical trials, we completed doses of FB2001 that were safe, and were projected to be effective in patients according to its pharmacokinetic profile.

This study is a double-blind, randomized, placebo-controlled study to evaluate the efficacy and safety of FB2001 in hospitalized patients with moderate to severe Coronavirus Disease 2019 (COVID 19). A total of about 1188 subjects are planned to be enrolled. The subjects will be randomized in a 1:1 ratio to FB2001 group or placebo group while both receiving standard of care treatment.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old, male or female.
2. Subjects hospitalized with moderate to severe COVID-19 with a category 4 or 5 on an 8-category ordinal scale.
3. Has laboratory-confirmed COVID-19 infection within 5 days prior to randomization.
4. Initial COVID-19 symptom onset within 5 days prior to randomization and ≥1 sign/symptom attributable to COVID-19 within 24 hours before randomization.
5. The underlying medical condition was well controlled prior to SARS CoV 2 infection and does not affect daily life.
6. Subject who did not receive COVID 19 (primary series or booster) vaccine within the 6 months prior to screening.
7. The subject is willing to provide written informed consent to participate in the study after reading the informed consent form and the information provided and has had the opportunity to discuss the study with the Investigator or designee.
8. The subject is able to communicate satisfactorily with the Investigator and to participate in, and comply with, the requirements of the study.
9. The subject is able to understand the nature of the study and any potential hazards associated with participating in it.
10. Negative pregnancy test for female subjects of childbearing potential and female subjects less than 2 years of postmenopause. Women of childbearing potential (WOCBP) and Women of non-childbearing potential are eligible to participate. Both women of childbearing potential and women of non-childbearing potential must use an approved method of birth control and agrees to continue to use this method for the duration of the study and for 30 days after taking the last dose of FB2001.

Exclusion Criteria:

1. Pregnant or breastfeeding, or intending to become pregnant during the study or within 30 days after the final dose or who are not willing to use a highly effective method of contraception.
2. HIV-infected subjects with viral load greater than 400 copies/mL or CD4 count less than 200 cell/µL from known medical history within past 6 months of the Screening Visit.
3. Subject with moderate to severe hepatic impairment or acute liver failure.
4. Known severe kidney disease.
5. Participated in other intervention studies within 6 months.
6. Has any condition for which, in the opinion of the Investigator, participation would not be in the best interest of the participant or that could prevent, limit, or confound the protocol-specified assessments including but not limited to participants who are not expected to survive longer than 48 hours after randomization, or participants who are expected to require mechanical ventilation within 48 hours after randomization, or participants with a recent history of mechanical ventilation.
7. Subjects receiving any medications or substances that are strong inhibitors or inducers of CYP3A within 14 days of randomization.
8. Received, ongoing or planed treatment with other anti-SARS CoV 2 therapeutics (including but not limited to known anti-SARS CoV 2 antibodies, small molecule antivirals, etc., other than remdesivir).
9. Other conditions that may increase the risk of study participation or, in the Investigator's judgment, make the participant inappropriate for the study.
10. Have known hypersensitivity to FB2001 or its excipients.
11. Any planned vaccine within 28 days following the last administration of FB2001 for Injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1188 (Estimated)
Dates: Start 2022-09-14 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Time to sustained recovery (in days) from randomization up to Day 29. | Up to Day 29
  Day of sustained recovery is defined as the first day on which a subject is discharged from hospital, or hospitalized for infection-control or other non-medical reasons through Day 29

SECONDARY OUTCOMES:
Proportion of participants with mechanical ventilation or all-cause-death | Through Day 29 and Day 60
  Proportion of participants with mechanical ventilation or all-cause-death in FB2001 group and placebo group
Proportion of participants with sustained recovery on Day 6 | On Day 6
  no specific description
Clinical status category as assessed by an 8-category ordinal scale daily while hospitalized and on Days, 15 and 29. | On Days 15 and 29
  no specific description
Duration of each targeted COVID-19 sign/symptom until discharge | Up to Day 29
  Duration of each targeted COVID-19 sign/symptom until discharge
Severity of each targeted COVID-19 sign/symptom until discharge | Up to Day 29
  no specific description
Days of supplemental oxygen (if applicable) | Up to Day 29
  no specific description
Duration of non-invasive ventilation/high-flow oxygen (if applicable) | Up to Day 29
  no specific description
Days of invasive mechanical ventilation/ECMO (if applicable) | Up to Day 29
  no specific description
Time to achieve SARS-CoV-2 virologic clearance | Up to Day 29
  no specific description
Proportion of participants achieving SARS-CoV-2 virologic clearance on Day 3, 5, 8, 15 and 29 | On Day 3, 5, 8, 15 and 29
  no specific description
Viral load change (log10) from baseline on Day 3, 5, 8 and 15. | On Day 3, 5, 8 and 15
  no specific description
Population pharmacokinetic (PK) parameters to be measured/analyzed, including AUC, Cmax and Ctrough | Day0-Day 5
  no specific descriptionsa

OTHER OUTCOMES:
Incidence and severity of Treatment-Emergent Adverse Events (TEAEs) | Up to Day 60
  safety evaluation
Incidence of withdrawals due to Adverse Events (AEs) | Up to Day 60
  safety evaluation
Incidence of Treatment-Related Adverse Events (TRAEs) | Up to Day 60
  safety evaluation
Incidence of Serious Adverse Events (SAEs) | Up to Day 60
  safety evaluation
Change/shifts in laboratory values from baseline | Up to Day 29
  safety evaluation
Change in vital signs including blood pressure, heart rate, respiratory rate, and temperature from baseline | Up to Day 29
  safety evaluation
Change in abnormal Electrocardiogram (ECG) parameters from baseline | Up to Day 29
  safety evaluation
Changes in abnormal physical examination findings from baseline | Up to Day 29
  safety evaluation
Change in oxygen saturation (SpO2) from baseline | Up to Day 29
  safety evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Yao, Study Director — Frontier Biotechnologies Inc.
Locations (2):
- China (2):
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Beijing Ditan Hospital Capital Medical University, Beijing

REFERENCES:
- [Derived] Shang W, Dai W, Yao C, Xu L, Tao X, Su H, Li J, Xie X, Xu Y, Hu M, Xie D, Jiang H, Zhang L, Liu H. In vitro and in vivo evaluation of the main protease inhibitor FB2001 against SARS-CoV-2. Antiviral Res. 2022 Dec;208:105450. doi: 10.1016/j.antiviral.2022.105450. Epub 2022 Oct 29. PMID 36354082